CLINICAL TRIAL: NCT00818090
Title: A Phase II Study of Paclitaxel and Cisplatin in Previously Untreated, Unresectable Invasive Thymoma or Thymic Carcinoma
Brief Title: Paclitaxel and Cisplatin for Thymic Neoplasm
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: marginal statistical significance
Sponsor: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Se-Hoon Lee, Korean Cancer Study Group, Korean Cancer Study Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-LU08-03; CRCST-L-0003
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2012-09

CONDITIONS: Thymoma; Thymic Carcinoma
Keywords: thymic epithelial tumor; paclitaxel; cisplatin; thymic carcinoma; invasive thymoma
MeSH Terms: conditions — Thymoma; Thymic epithelial tumor | interventions — TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TP (Experimental): paclitaxel and cisplatin every 3 weeks
  Interventions: Drug: paclitaxel and cisplatin

INTERVENTIONS:
Drug: paclitaxel and cisplatin — paclitaxel and cisplatin every 3 weeks

SUMMARY:
To assess the efficacy and safety of the regimen in previously untreated, unresectable invasive thymoma or thymic carcinoma

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed invasive thymoma or thymic carcinoma
* unresectable tumor: by either local invasion, distant metastasis, or recurred (assessed by investigator)
* no previous systemic treatment for invasive thymoma or thymic carcinoma
* at least one measurable lesion by RECIST criteria
* 18 years old or older
* ECOG performance status 0, 1, 2
* adequate lab. findings neutrophil ≥ 1.5 x 10^9/L platelet ≥ 75 x 10^9/L hemoglobin ≥ 9.0 g/dL bilirubin ≤ 1.5 x upper normal limit AST, ALT ≤ 2.5 x upper normal limit Alkaline phosphatase ≤ 2.5 x upper normal limit (if liver metastasis, ≤ 5 x upper normal limit) serum creatinine ≤ 1.0 x upper normal limit if serum creatinine > 1.0 x upper normal limit, creatinine clearance ≥ 60 mL/min
* patient who agree to written, informed consent

Exclusion Criteria:

* other malignancy (exception: non-melanoma skin cancer, cervical carcinoma in situ, cancer without evidence more than 5 years since curative resection)
* active bacterial infection
* history of clinical trial with investigational drug within 30 days
* radiotherapy to thoracic or mediastinal area (other area radiotherapy is permitted)
* pregnant, or lactating women
* patient with organ transplantation
* peripheral neuropathy, grade 2 or greater
* severe, medical condition unstable cardiac disease despite of adequate management myocardial infarction within 6 months active ulcer disease refractory to medication chronic obstructive lung disease requiring admission treatment within 1 year
* uncontrolled seizure, cerebral nervous system disorder, psychiatric problem which decrease treatment compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 weeks, 12 weeks, 18 weeks

SECONDARY OUTCOMES:
toxicity | start of medication to 4 weeks since the last medication
progression-free survival | till progression
duration of response | till progression
overall survival | till death, last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dae Seog Heo, MD, PhD, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea